CLINICAL TRIAL: NCT00211068
Title: Retrospective Case-control Study of Risk Factors for Anti-erythropoietin Antibody Positive Pure Red Cell Aplasia Among Patients With Chronic Kidney Disease Receiving Epoetin Alfa
Brief Title: A Study of Risk Factors for Anti-erythropoietin Antibody Positive Pure Red Cell Aplasia Among Patients With Chronic Kidney Disease Receiving Epoetin Alfa
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004408; EPO-IMU-403 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Pure Red-cell Aplasia
Keywords: Pure red-cell aplasia; Chronic kidney failure; Epoetin alfa (Eprex); Erythropoietin; Kidney disease; Anemia
MeSH Terms: conditions — Red-Cell Aplasia, Pure; Kidney Failure, Chronic; Kidney Diseases; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood sample collected for pharmacogenomic analysis
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Epoetin alfa: Four control patients will be matched to each index patients enrolled in protocol EPO-IMU-301 identified as having chronic kidney disease and an immune-mediated cause of pure red cell aplasia (PRCA) indicated by the presence of anti-erythropoietin (EPO) antibodies in their serum at the time of loss of efficacy.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This study is an observational study. No medication will be provided or administered to the participants. Participants will receive standard-of-care treatment from their individual physicians.
  Other Names: EPREX

SUMMARY:
The purpose of this study is to collect historical occurrences of risk factors that are potentially associated with the development of anti-erythropoietin (EPO) antibody positive pure red cell aplasia (PRCA) in participants with chronic kidney disease who have been recently treated with epoetin alfa (EPREX).

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), case-control (study that compare individuals with a disease or condition [cases] to a group of individuals without the disease or condition [controls] to determine the possible factor which increased disease incidence), retrospective (a study in which the participants are identified and then followed backward, as time passes) study. Retrospective risk factor data will be collected for control participants matched to the subset of participants in Protocol EPO-IMU-301 identified as having chronic kidney disease and anti-EPO antibody positive PRCA that began while the participant was receiving treatment with EPREX (index participants). For each index participant, up to 4 matched non-PRCA control participants with chronic kidney disease will be enrolled in this study. Approximately 600 control participants will be enrolled in this study. Control participants will be selected from the same site as the index participant and the data will be collected from the date closest to the reference date (loss of efficacy [drop in hemoglobin of greater than 2 g/dL/month] was first seen) that the control participant satisfies all study inclusion and exclusion criteria. The optional pharmacogenomic part (testing for polymorphisms and haploid types of the erythropoietin gene) will be recorded for the control participants who will sign the pharmacogenomics part of the study. No drug administration or treatment will be mandated by this study. Safety evaluation will include assessment of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* History of anemia due to chronic kidney disease
* Pure red cell aplasia (PRCA) associated with erythropoietin-alpha (EPO) treatment
* Treatment with EPO for a minimum of 2 months occurring within more or less 3 months of the reference date (date of loss of efficacy [drop in hemoglobin of greater than 2 g/dL/month] was first observed)

Exclusion criteria

* History of and information related to past exposure to EPO not available
* History of PRCA or anti-EPO antibody positive status before or after the reference date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants having chronic kidney disease and an immune-mediated cause of pure red cell aplasia indicated by the presence of anti-erythropoietin antibodies in their serum at the time of loss of efficacy
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2004-03; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Study medication-related risk factors: Number of participants who received Human Serum Albumin (HSA) containing drug | 1 year prior to the reference date
  The reference date is the day on which Loss of Efficacy (LOE) was first suspected, where LOE is the date that a drop in hemoglobin of greater than 2 g/dL/month was first seen.
Study medication-related risk factors: Number of participants who received HSA-free drug | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants who received epoetin alfa intravenously | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants who received epoetin alfa subcutaneously | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants who self-administered epoetin alfa | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants who administered epoetin alfa in hospital or in clinic | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants with the duration of epoetin alfa treatment | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants with the duration of other recombinant human erythropoietins (r-HuEPOs) treatment | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants with exposure to epoetin alfa | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants with exposure to other r-HuEPOs | 1 year prior to the reference date
Study medication administration-related risk factors: Number of participants with frequency of epoetin alfa dosing | 6 months prior to the reference date
Study medication administration-related risk factors: Number of participants with frequency of other r-HuEPOs dosing | 6 months prior to the reference date
Participant-related risk factors: Number of participants according to age | 1 year prior to the reference date
Participant-related risk factors: Number of participants according to sex | 1 year prior to the reference date
Participant-related risk factors: Number of participants according to race | 1 year prior to the reference date
Participant-related risk factors: Number of participants according to underlying diagnosis of chronic kidney disease | 1 year prior to the reference date
Participant-related risk factors: Number of participants according to type of renal replacement therapy (if any at the time of the reference date) | 1 year prior to the reference date
Participant-related risk factors: Number of participants with history of malnutrition | 1 year prior to the reference date
Participant-related risk factors: Number of participants with history of autoimmune disease or positive results of autoimmune testing | 1 year prior to the reference date
Participant-related risk factors: Number of participants with history of immune dysregulation | 1 year prior to the reference date
Participant-related risk factors: Number of participants with uncontrolled hyperparathyroidism | 1 year prior to the reference date
Participant-related risk factors: Number of participants with uncontrolled hypothyroidism | 1 year prior to the reference date
Participant-related risk factors: Number of participants with history of malignancy | 5 years prior to the reference date
Participant-related risk factors: Number of participants with history of viral infection | 1 year prior to the reference date
Participant-related risk factors: Number of participants with history of vaccination | 1 year prior to the reference date
Participant-related risk factors: Number of participants with immunosuppressive/immunomodulatory therapy | 1 year prior to the reference date
Participant-related risk factors: Number of participants with history of frequent transfusions | 1 year prior to the reference date
Participant-related risk factors: Number of participants with treatment with other subcutaneous medications | 1 year prior to the reference date
Participant-related risk factors: Number of participants with treatment with other recombinant human proteins | 1 year prior to the reference date
Participant-related risk factors: Number of participants who received other concomitant therapy | 1 year prior to the reference date

SECONDARY OUTCOMES:
Human leukocyte antigen (HLA) typing | 1 year prior to the reference date
  The optional pharmacogenomic (use of genetic information to predict whether the study medication will help make a patient well or ill) part of the study will test for polymorphisms and haploid types of the erythropoietin gene. HLA typing will be recorded for the control participants who will sign the pharmacogenomics part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L. L. C. Clinical trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (22):
- Brazil (2):
  - São Paulo
  - Sorocaba
- France (5):
  - Bois-Guillaume
  - Grenoble
  - Nantes
  - Orléans
  - Paris
- Tvnsberg, Norway
- Bloemfontein, South Africa
- Sweden (3):
  - Karlshamn
  - Stockholm
  - Trollhättan
- Vlissingen, Thailand
- United Kingdom (9):
  - Birmingham
  - Brighton
  - Bristol
  - Chelmsford
  - Edinburgh
  - London
  - Manchester
  - Omagh
  - Westcliff-on-Sea